CLINICAL TRIAL: NCT06661655
Title: Evaluation of a New Ultrasound System for the Non-invasive Assessment of Liver Steatosis in MASLD/MASH Patients
Acronym: ACOUSTIQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: E-Scopics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ES213; 2023-A02456-39 (Other: French ANSM)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Syndrome X; Fatty Liver; MASH - Metabolic Dysfunction-Associated Steatohepatitis; MASLD; NASH (Non-Alcoholic Steatohepatitis); Steatosis, Liver; NAFLD
Keywords: Liver; Fibrosis; Steatosis; Elastography; Ultrasound; Attenuation; Backscattering coefficient; Sound speed; MRI PDFF; Hepatoscope
MeSH Terms: conditions — Metabolic Syndrome; Fatty Liver; Non-alcoholic Fatty Liver Disease; Fibrosis

STUDY DESIGN:
Intervention Model Description: Cross sectional investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main cohort (Experimental): Patients recruited in the study will receive an ultrasound exam with Hepatoscope to collect quantitative measurements related to the severity of liver steatosis.
  Interventions: Device: Liver ultrasound

INTERVENTIONS:
Device: Liver ultrasound — Hepatoscope is a point of care ultraportable ultrasound device that is capable of conventional grayscale ultrasound imaging, of 2D transient elastography (imaging + liver stiffness measurement), and of quantitative ultrasound properties measurement (ultrasound attenuation, backscattering coefficient, sound speed) related to liver steatosis.

SUMMARY:
The objective of the study is to evaluate an ultraportable ultrasound device, Hepatoscope, for the non-invasive assessment of hepatic steatosis in patients with metabolic-dysfunction associated liver diseases (MASLD), by comparing its measurements with current diagnostic modalities, such as MRI-PDFF.

DETAILED DESCRIPTION:
The objective of the study is to evaluate an ultraportable ultrasound device, Hepatoscope, for the non-invasive assessment of hepatic steatosis in patients metabolic-dysfunction associated liver diseases (MASLD), by comparing its measurements with current diagnostic modalities, such as MRI PDFF.

The primary objective is to compare ultrasound parameters measurements of ultrasound attenuation, backscattering coefficient and sound speed to the hepatic fat fraction as measured with MRI-PDFF.

The secondary objectives includes the comparison of measurements of quantitative ultrasound parameters between Hepatoscope and FibroScan, and to compare the measurement of liver stiffness between Hepatoscope and MRE.

Exploratory objectives have been determined to allow the comparison of said measured parameters to the outcome of histopathological analysis in a subset patient population who would benefit from a liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient below 80 yo
* Patients with MASLD/MASH recruited in interventional trials requiring MRI PDFF +/- MRE per interventional protocol, OR
* Patients with MASLD/MASH recruited in prospective cohorts requiring MRI PDFF +/- MRE per interventional protocol, OR
* Patients referred to MRI-PDFF or MRE.
* Patients who consented in written to participate in the study
* Patients with ongoing social security coverage

Exclusion Criteria:

* Patient in their minority (less than 18 yo) or older than 80 yo,
* Patient with active implants,
* Patient presenting with a wound where the Hepatoscope exam shall be performed (abdominal right upper quadrant)
* Patient with a history of decompensated cirrhosis,
* Patient with a history of hepatocellular carcinoma,
* Adult patient under tutorship, or unable to express informed consent,
* Pregnant or breast-feeding
* Person deprived from their liberty
* Patient hospitalized without providing consent or in case of an emergency
* Patient presenting with another know liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation with MRI PDFF | At a maximum of 6 months from enrollment
  Spearman correlation coefficients between each Hepatoscope measurement (ATT, BSC and SOS) and MRI-PDFF measurements will be calculated. The confidence interval will be estimated with an alpha risk of 0,017 (Bonferroni adjustment, overal alpha risk of 0,05). Each correlation will be compared to the lowest acceptable threshold D = 0,50 with a Fisher Z test, with an alpha risk de 0,017.

SECONDARY OUTCOMES:
Comparison with Fibroscan CAP | At a maximum of 6 months from enrollment
  Spearman correlations between Hepatoscope measurements and MRI-PDFF will be compared to Spearman correlations between Fibroscan CAP measurements and MRI-PDFF. The 95% confidence interval of each correlation will be estimated and compared to each other using a Fisher Z test with an alpha risk of 0,05.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Cohen-Bacrie, Study Director — E-Scopics; Jerome Boursier, MD, PhD, Study Chair — University Hospital, Angers
Locations (3):
- France (3):
  - University Hospital Angers, Angers
  - Beaujon University Hospital, Clichy
  - Pitie Salpetriere University Hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified individual participant data may be shared, limited to data collected in CRF